CLINICAL TRIAL: NCT00693446
Title: An Open-Label, Comparative, Randomized, Prospective Study To Compare Sirolimus Versus Tacrolimus In De Novo Simultaneous Pancreas- Kidney Allograft Recipients Receiving An Induction Therapy With Antithymocyte Globulin Plus Mycophenolate Mofetil Plus Corticosteroids
Brief Title: A Study To Compare Sirolimus Versus Tacrolimus In De Novo Simultaneous Pancreas- Kidney Allograft Recipients Receiving An Induction Therapy With Antithymocyte Globulin Plus Mycophenolate Mofetil Plus Corticosteroids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/04/2-D
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Pancreas Transplantation; Kidney Transplantation
Keywords: Pancreas-kidney allograft; tacrolimus; sirolimus; Pancreas-kidney allograft recipients
MeSH Terms: interventions — Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): In a first period, the patient will receive Tacrolimus. The time of first administration will be within the first 48H post transplantation.
  In a second period, the patient will receive Sirolimus. The time of first administration of Sirolimus will be between day 60 and day 90 post transplant. Tacrolimus will be stopped at that time.
  Interventions: Drug: Sirolimus
- 1 (Other): Patients receive Tacrolimus from day 0 to the end of the study (Arm Tacrolimus).
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Sirolimus — In a first period, the patient will receive Tacrolimus. The time of first administration will be within the first 48H post transplantation. The initial dose will be 0,1 mg/day po. then titrated to maintain trough whole-blood concentrations between 5-15 ng/ml.
  In a second period, the patient will receive Sirolimus. The time of first administration of Sirolimus will be between day 60 and day 90 post transplant. Tacrolimus will be stopped at that time.
  The initial dose will be 8 mg/day po. till a trough level is obtained and then titrated to maintain trough whole-blood concentrations between 5-15ng/ml.
  The dose of sirolimus will be administrated once a day.
  Arms: 2
Drug: Tacrolimus — Patients receive Tacrolimus from day 0 to the end of the study. The time of first administration will be within the first 48 hours post transplant.
  The dose of tacrolimus will be administrated twice a day. The initial dose will be 0,1 mg/day po. then titrated to maintain trough whole-blood concentrations between 5-15 ng/ml.
  Patients receive also rATG , mycophenolate mofetil and corticosteroids.
  Arms: 1

SUMMARY:
Experience with tacrolimus in pancreas transplantation has become a standard for immunosuppression in almost all pancreas centers over the world. Several centers have shown very good results in simultaneous pancreas-kidney (SPK) transplant recipients receiving antithymocyte globulin induction and maintenance immunosuppression consisting of calcineurin inhibitor and mycophenolate mofetil with or without corticosteroids.

The use of sirolimus in SPK transplant patients has for the moment only been studied, with good results, in association with tacrolimus or cyclospsorine (CsA). In renal transplantation, there is also evidence that sirolimus (Rapamune) is a potent immunosuppressant that significantly reduces the incidence of acute rejection when given with CsA, effective as base therapy in the post-induction period. Because of Rapamune's effectiveness and different safety profile, it might be advantageous in terms of reduced nephrotoxicity to avoid completely calcineurin inhibitors without increased incidence of acute rejection.

To explore this further, the following study is designed to assess the use of SRL versus TAC, both treatment groups including rATG plus MMF and a 3-month course of steroids in de novo simultaneous pancreas-kidney transplant recipients.

DETAILED DESCRIPTION:
The main objective is to compare renal and pancreas graft survivals at 12 months after simultaneous pancreas-kidney transplantation in patients receiving either a regimen combining sirolimus (SRL) plus mycophenolate mofetil (MMF) following an antibody induction (rATG) or a regimen combining tacrolimus (TAC) plus mycophenolate mofetil following an antibody induction (rATG). In both regimens corticosteroids (CS) will be withdrawn three months after transplantation.

In addition, the two treatment groups will be compared for acute rejection, renal and pancreas functions and patient survival after transplantation at 12 months and for a total period of 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age ≥ 18 and ≤ 60 years.
* Patients receiving a first cadaveric simultaneous pancreas-kidney transplant for insulin-dependent diabetes associated with end-stage renal disease.
* Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation.
* Signed and dated informed consent.

Exclusion Criteria:

* Donor age ≤ 15 years and ≥ 60 years.
* Evidence of active systemic or localized major infection.
* Evidence of infiltrate, cavitation, or consolidation on chest x-ray.
* Use of any investigational drug or treatment (in particular immuno-suppressive drugs) up to 4 weeks prior to enrollment to the study and during the 12-month treatment phase.
* History of malignancy (with the exception of adequately treated localized squamous cell or basal cell carcinoma, without recurrence within 5 years of enrolment into the study).
* Graft from a living donor.
* Double renal graft.
* Pregnancy.
* Known hypersensitivity to sirolimus and its derivatives or to tacrolimus.
* Known hypersensitivity to rabbit's proteins.
* Multiple organ transplants or recipients of previously transplanted organs other than kidney.
* Treatment with cisapride (PrépulsidÒ), pimozide (OrapÒ), ketoconazole (NizoralÒ), fluconazole (TriflucanÒ) or millepertuis (ProcalmilÒ, Arkogélules MillepertuisÒ), that is not discontinued within 24 hours prior to transplant.
* Total white blood cell count ≤ 2 x 109/L or platelet count ≤ 70.000/mm3 at baseline.
* Patients with evidence of active histological or biological hepatic disease during the six months period before the transplantation.
* HIV positive recipients.
* Non-heart beating donor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2004-04; Primary Completion 2013-04 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Kidney graft and pancreas graft survivals at month 12. | 12 months

SECONDARY OUTCOMES:
Incidence of histologically proven acute rejection episode at 3, 6, 12 months then annually up to 60 months. | 60 months
Incidence of presumed clinical acute rejection at 3, 6, 12 months then annually up to 60 months. | 60 months
Incidence of patient survival at 12 months then annually up to 60 months. | 60 months
Incidence of renal graft survival annually up to 60 months. | 60 months
Incidence of pancreas graft survival annually up to 60 months. | 60 months
Time to the first acute rejection episode (time to the beginning of treatment of acute rejection episode).
Severity of rejection episodes including a histological grade of the first acute rejection episode.
Incidence of documented infection (culture, biopsy or serologically confirmed) or presumptive infection, including opportunistic infections at 3, 6, 12 months then annually up to 60 months. | 60 months
Incidence of histologically-confirmed lymphoproliferative disease or malignancy at 12 months then annually up to 60 months. | 60 months
Renal function assessed by creatinine clearance (Cockroft and Gault's formula) at 3, 6 and 12 months then annually up to 60 months. | 60 months
Renal function assessed by serum creatinine at 3, 6 and 12 months then annually up to 60 months. | 60 months
Incidence of renal Delayed Graft Function (DGF) defined as the need for more than one dialysis during the first week following transplantation.
Duration of renal Delayed Graft Function.
Incidence of renal Slow Graft Function (SGF) defined as serum creatinine ≥ 250 µmol/l at day 5 after transplantation (in the absence of dialysis).
Histology of renal graft will be assessed at month 12 if biopsy is not contra-indicated. | At month 12
Pancreas graft function evaluated by hemoglobin A1C (HbA1C) at 3, 6 and 12 months then annually up to 60 months. | 60 months
Pancreas graft function evaluated by basal glycemia at 3, 6 and 12 months then annually up to 60 months. | 60 months
Pancreas graft function evaluated by stimulated glycemia levels at 6 and 12 months then annually up to 60 months. | 60 months
Pancreas graft function evaluated by basal insulin secretion at 3, 6 and 12 months then annually up to 60 months. | 60 months
Pancreas graft function evaluated by stimulated insulin secretion at 6 and 12 months then annually up to 60 months. | 60 months
Incidence of hypertension (defined as systolic ≥ 140 mmgHG and/or diastolic ≥ 90 mmgHG and the use of antihypertensive medications including diuretics) at 3, 6 and 12 months then annually up to 60 months. | 60 months
Number of antihypertensive drugs at 3, 6 and 12 months then annually up to 60 months. | 60 months
Lipid levels (cholesterol, triglycerides, LDL-cholesterol, HDL-cholesterol) at 3, 6 and 12 months then annually up to 60 months. | 60 months
Number of lipid lowering agents at 3, 6 and 12 months then annually up to 60 months. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Diego CANTAROVICH, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, Nantes, France

REFERENCES:
- [Derived] Cantarovich D, Kervella D, Karam G, Dantal J, Blancho G, Giral M, Garandeau C, Houzet A, Ville S, Branchereau J, Delbos F, Guillot-Gueguen C, Volteau C, Leroy M, Renaudin K, Soulillou JP, Hourmant M. Tacrolimus- versus sirolimus-based immunosuppression after simultaneous pancreas and kidney transplantation: 5-year results of a randomized trial. Am J Transplant. 2020 Jun;20(6):1679-1690. doi: 10.1111/ajt.15809. Epub 2020 Feb 28. PMID 32022990